CLINICAL TRIAL: NCT01551576
Title: Photoacoustic Imaging (PAI) of the Prostate: A Clinical Feasibility Study
Status: Completed | Type: Observational
Sponsor: Stanford University (Other)
Responsible Party: Sponsor
Other Study IDs: IRB-22701; SU-03012012-9209 (Other: Stanford University); PROS0046 (Other: OnCore)
Record Dates: First submitted 2012-03-08; First posted 2012-03-12 (Estimated); Last update posted 2021-11-02 (Actual); Status verified 2021-10

CONDITIONS: Prostate Cancer
MeSH Terms: conditions — Prostatic Neoplasms

STUDY DESIGN:
Observational Model: Other | Time Perspective: Cross-Sectional
Oversight: Data Monitoring Committee: Yes | FDA-regulated Drug: No | FDA-regulated Device: No | US Export: No

GROUPS / COHORTS (1):
- photoacoustic imaging (PAI): Men seen in the urology clinic for elevated PSA and/or abnormal digital rectal exam (DRE) will be offered PAI at the time of transrectal ultrasound guided biopsy, which is standard of care. In addition, patients with a biopsy proven prostate cancer may also be approached for this PAI scan
  Interventions: Device: Hand held transrectal Combined Ultrasound and photoacoustic imaging (PAI) probe

INTERVENTIONS:
Device: Hand held transrectal Combined Ultrasound and photoacoustic imaging (PAI) probe — Hand held transrectal Combined Ultrasound and photoacoustic imaging (PAI) probe. PAI is a non-ionizing imaging technique

SUMMARY:
The purpose of our study is to image human prostate tissue using a transrectal photoacoustic imaging probe.

DETAILED DESCRIPTION:
PRIMARY OBJECTIVE(S):

The primary objective of this pilot study is to assess PAI-performance in a clinical setting to understand limitations of our current PAI instrumentation and to help improve the next-generation design.

SECONDARY OBJECTIVE(S):

To do preliminary evaluations of oxygen saturation in lesions based on PAI-measurements in order to distinguish malignant from benign prostatic tissue as a basis for future studies.

ELIGIBILITY:
Inclusion Criteria:

* Consent signed
* Male >= 18 and <= 80 years of age
* Patients must have an elevated PSA And/ Or Abnormal digital rectal exam Or Other indication for prostate biopsy Or Patients with biopsy proven prostate cancer who are scheduled for prostatectomy.

Exclusion Criteria:

* History of prostatectomy or other surgical history that would preclude transrectal imaging (i.e. abdominal perineal resection), anal stenosis/stricture disease
* Men with anatomic abnormalities or previous surgical history that make transrectal imaging impossible (for example, men with previous abdominal-perineal bowel resections or anal atresia/stenosis)

Ages: 18 Years to 80 Years | Sex: Male | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Study Population: Medical oncologists with appropriate patient populations will be informed of the study and the inclusion and exclusion criteria. Potential participants will be recruited from the Stanford Urologic Oncology Clinic. A study investigator will follow-up with participants who are interested in participating in this study. Study information will be posted on the Stanford Cancer Center website as well.
Sampling Method: Non-Probability Sample
Enrollment: 20 (Actual)
Dates: Start 2014-02 (Actual); Primary Completion 2019-12-16 (Actual); Study Completion 2019-12-16 (Actual)

PRIMARY OUTCOMES:
lesion signal intensity on Photoacoustic Imaging (PAI) in relation to different lesion characteristics and the surrounding tissues | 36 months
  measure of the lesion signal intensity on PAI in relation to different lesion characteristics and the surrounding tissues. The average signal intensity (or more specifically the SNR) of the lesions measured in dB) will be tabulated against lesion depth from the transducer, and lesion size, based on ultrasound measurements

SECONDARY OUTCOMES:
Measures of hypoxia in the lesion | 36 months
  total lesion hemoglobin concentration (HbT) at PAI and percentage SO2 (oxygen saturation) in region of interest (ROI) (average and maximum) which will be tested against lesion characteristics based on histology at pathological examination of the biopsy and/or prostatectomy specimen if the patients proceed to have radical prostatectomy performed

CONTACTS AND LOCATIONS:
Overall Officials: Andrei H Iagaru, MD, PhD, Principal Investigator — Stanford University; Martin Karl Schneider, PhD, Principal Investigator — Stanford University
Locations (1):
- Stanford University Cancer Institute, Stanford, California, United States

IPD SHARING:
Plan to Share IPD: No